CLINICAL TRIAL: NCT06673615
Title: A Community-based Cohort Study on Early Screening of Heart Failure in Elderly Population in Shanghai
Brief Title: A Cohort Study on Early Stages of Heart Failure
Status: Recruiting | Type: Observational
Sponsor: Shanghai East Hospital (Other)
Collaborators: Beicai Community Health Service Center of Pudong District, Shanghai, China (Unknown)
Responsible Party: Sponsor
Other Study IDs: XSDL-001
Record Dates: First submitted 2024-09-23; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Stages of Heart Failure
Keywords: Heart failure; Early screening; Elderly population; Epidemiology
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Stages of Heart Failure in a Community-based Cohort China: A community-based cohort on stage A (at risk for HF), stage B (pre-HF) or stage C (symptomatic HF) of heart failure in China elderly people

SUMMARY:
The main goal of this observational study is to learn about the epidemiological characteristics of heart failure among elder population in Beicai community in Shanghai and construct a community-based database and biobank. The main question it aims to answer is:

What is the prevalence and prognosis of different stages of heart failure among elder population in community in Shanghai? And what are the influencing factors? What are the best screening strategies and hierarchical management strategies among different stages of heart failure patients in community? Participants are the elderly people aged 60 years or older in Beicai community in China. The follow-up will be programmed every 2 years.

DETAILED DESCRIPTION:
Heart failure is a serious manifestation or advanced stage of various heart diseases with high mortality and re-hospitalization rates, and early diagnosis of heart failure is important to improve patient survival. Currently, the prevalence of preclinical heart failure (heart failure stage B) is lacking in China, and the rate of progression of heart failure from stage A/B to symptomatic heart failure (heart failure stage C) and end-stage heart failure (heart failure stage D) and the factors influencing the heart failure development are unknown.

The study is an ongoing prospective community-based study. After enrollment, a questionnaire, physical examination, laboratory examination and imaging examination will be administered to each participant at baseline and every 2 years in the follow-up. The laboratory and imaging examination include: blood/urine sample and biochemical measurements, electrocardiogram, echocardiograph, etc. In the follow-up, the incidence of cardiovascular disease, heart failure, other CV events and mortality will be recorded. Whether at baseline or follow-up, if the investigators find that patients are unclear about their disease status, the investigators will notify them by phone and record their subsequent medical behavior and results.

In this study, a community-based database and biobank will be established for early screening and long-term prognosis of heart failure in elderly population. Through the analysis of the data, the epidemiological characteristics of early stage of heart failure in elderly population in Shanghai can be identified and a multivariable model predicting heart failure in early stage will be constructed. Furtherly，the investigators will explore the referral criteria and hierarchical management strategies for heart failure through the cooperation between community hospitals and comprehensive hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥60 years
2. Cooperate in participating in research and sign informed consent forms

Exclusion Criteria:

1. End stage heart failure patients
2. Refusal to participate in this study
3. Patients who are not suitable to participate in this study by Researchers's evaluation

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly people who have signed informed consent forms for physical examinations in Beicai Community
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2034-08-30 (Estimated); Study Completion 2044-08-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality rate | 10 years
  All-cause mortality rate of different stages of heart failure

SECONDARY OUTCOMES:
Prevalence of early heart failure | 10 years
  The prevalence of early heart failure was defined as morbidity of stage A heart failure and stage B heart failure. Stage A HF was defined as at risk for HF but without current or previous symptoms/signs of HF and without structural/functional heart disease or abnormal biomarkers.(eg. patients with hypertension, coronary artery disease, diabetes, obesity, atrial fibrillation/atrial flutter or tumour). Stage B HF was defined as no symptoms or signs of HF and evidence of one of the following:1) EF value<52 in male and <54 in female. 2) Increased NT-proBNP levels (≥125 pg/ml) or elevated TnT levels (>0.017ng/ml).
Progress of heart failure of Stage A | Following up 10 years
  The morbidity rate of stage B heart failure, stage C heart failure and stage D heart failure in stage A heart failure patients in 2 year, 6 years and 10 years. Stage A HF was defined as at risk for HF but without current or previous symptoms/signs of HF and without structural/functional heart disease or abnormal biomarkers.(eg. patients with hypertension, coronary artery disease, diabetes, obesity, atrial fibrillation/atrial flutter or tumour). Stage B HF was defined as no symptoms or signs of HF and evidence of one of the following:1)EF value<52 in male and <54 in female.2) Increased NT-proBNP levels (≥125 pg/ml) or elevated TnT levels (>0.017ng/ml). Stage C/D HF was defined as previous history of HF or structural heart disease with current or previous symptoms of HF (eg. dyspnea, swelling of both lower extremities), diagnosed by two cardiac specialists.
Progress of heart failure of Stage B | Following up 10 years
  The morbidity rate of stage C heart failure and stage D heart failure in stage B heart failure patients in 2 year, 6 years and 10 years. Stage B HF was defined as no symptoms or signs of HF and evidence of one of the following:1)EF value<52 in male and <54 in female.2) Increased NT-proBNP levels (≥125 pg/ml) or elevated TnT levels (>0.017ng/ml). Stage C/D HF was defined as previous history of HF or structural heart disease with current or previous symptoms of HF (eg. dyspnea, swelling of both lower extremities), diagnosed by two cardiac specialists.
Progress of heart failure of Stage C | Following up 10 years
  The morbidity rate of stage D heart failure in stage C heart failure patients in 2 year, 6 years and 10 years. Stage C HF was defined as previous history of HF or structural heart disease with current or previous symptoms of HF (eg. dyspnea, swelling of both lower extremities). Stage D HF was defined as Marked HF symptoms that interfere with daily life and with recurrent hospitalizations despite attempts to optimize GDMT.
Clinical endpoints of heart failure | Following up 10 years
  Time of first occurrence of symptomatic heart failure. Symptomatic heart failure was defined as current or previous symptoms/signs of HF.
New cardiovascular events | Following up 10 years
  Incidence rate of cardiovascular events
Referral rate | 10 years
  Proportion of patients referred to higher-level hospitals due to heart failure
Cardiovascular mortality rate | 10 years
  Cardiovascular mortality rate of different stages of heart failure

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gong X, Xu J, Wang M, Hu H, Yan Y, Han W, Huang J. Implementing community-based heart failure screening in primary care settings: a population-based pilot study in Shanghai, China. BMC Prim Care. 2025 Dec 18. doi: 10.1186/s12875-025-03124-1. Online ahead of print. PMID 41408608